CLINICAL TRIAL: NCT00636753
Title: Antipsychotics and Metabolic Syndrome
Status: Suspended | Type: Observational
Why Stopped: this study has not finding place
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: dr.med., centerchef Henrik Lublin, Psychiatric Center Glostrup
Other Study IDs: HC-2007-0070
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic and endocrine changes in schizophrenic patients by antipsychotics treatment.
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — whole blood, serum/plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: schizophrenic patients
- 2: controls

SUMMARY:
The purpose of the study is to determine whether antipsychotic treatment is influence psychiatric patients due to endocrine and metabolic status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Gender male
* Age 18-45
* Debut drug-naive schizophrenics,
* Caucasians
* Consent given to take part in the project

Exclusion Criteria:

* Compliance-problems
* Major lung-/kidney/hart/lever disorders
* Abuse of alcohol/drugs
* Diabetes 1 and 2
* Antihypertensive
* Anticholesterol-reducing medication
* Patients under duress

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with debut of schizophrenia, controls from database
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Psychiatric Center Glostrup, Copenhagen, Nordre Ringvej 28-69, Glostrup
  - Psychiatric Center Glostrup, Nordre Ringvej 28-69, Glostrup